CLINICAL TRIAL: NCT01771393
Title: Performance of Cone-beam Computed Tomography (CT) Compared to Multidetector CT for Arthrography of the Wrist, Ankle, Elbow and Knee
Brief Title: Cone-beam vs Multidetector Computed Tomography (CT) for Arthrography of the Wrist, Ankle, Elbow and Knee
Acronym: ARCOBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012.711
Record Dates: First submitted 2012-10-18; First posted 2013-01-18 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cartilage Ulceration of the Distal Joints
Keywords: arthroscanner; cone-beam computed tomodensitometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBCT prior to MDCT (Experimental): To avoid systematic bias in performance or image quality due to dilution of the contrast enhancement within the joint, the order of the CBCT and the MDCT will be randomized. This arm is composed of patients who will have the CBCT performed prior to the MDCT.
  Interventions: Device: CBCT prior to MDCT
- MDCT prior to CBCT (Experimental): To avoid systematic bias in performance or image quality due to dilution of the contrast enhancement within the joint, the order of the CBCT and the MDCT will be randomized. This arm is composed of patients who will have the MDCT performed prior to the CBCT.
  Interventions: Device: MDCT prior to CBCT

INTERVENTIONS:
Device: CBCT prior to MDCT — Cone-beam scanner is performed immediately after arthrography, then multidetector scanner is performed.
  Arms: CBCT prior to MDCT
Device: MDCT prior to CBCT — Multidetector scanner is performed immediately after arthrography, then Cone-beam scanner is performed.
  Arms: MDCT prior to CBCT

SUMMARY:
ConeBeam scanner (CBCT) is a widely technique used for dental and maxillofacial imaging. Patients can be set up in a sitting or a laying position in the, Newtom 5G CBCT allowing for an analysis of the limbs distal joints. Our hypothesis is that the cone-beam scanner could detect and characterize chondral lesions the cartilage similarly to a multidetector CT (MDCT). 100 patients over 18 years requiring arthroscanner of the wrist, ankle, elbow or knee will be enrolled The primary endpoint based on the ability of cone-beam scanner to detect cartilage lesions. Secondary endpoints will concern the depiction of the joint lesions, quality of the images, tolerability of the exams and inter- intra-operator reproducibility. After arthrography, patients will have a MDCT considered as the reference exam, and a CBCT on a randomized order. Exams will be anonymized and read twice by two trained radiologists with 3-6 week intervals. The inter-observer agreement for the diagnosis of cartilage lesion type between the two techniques will be evaluated by a kappa coefficient. The evaluation of diagnostic performance will be achieved by studying the sensitivity, specificity, negative predictive value and positive predictive value, and its likelihood ratio. Kappa test will be performed to evaluate the consistency of the depiction of the lesions. A Student t test will be performed for paired data if distributions are normal, a Wilcoxon test if not. To assess patient's tolerance, the percentages of (painful, not painful) will be calculated for each technique and will be compared using the Chi2 test (or Fisher's exact test if the chi can not apply).

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 years old or above, weight ≤ 160 Kg
* Patient require knee or ankle or elbow or wrist arthroscanner
* French spoken an read
* Free and informed consent signed
* Being affiliated to a French social security system or similar.

Exclusion Criteria:

* Patients already included in the ARCOBE study
* Patient with severe pain and reduced spontaneous mobility that could prevent proper positioning for the cone-beam
* Lack of effective contraception (risk of pregnancy) or pregnancy proven data on interrogations
* Patient on protection of the court, under supervision or trusteeship
* Inability to express a consent
* Patients already enrolled in a study with a conflict of interest with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
cartilage damage thickness | participants will be followed for the duration of the arthrography CT , an expected average of 2 hours
  0- normal, 1- Linear cartilage tear, 2- focal ulceration of less than 50% of the cartilage thickness, 3-: - focal ulceration of greater than 50% of the cartilage thickness, 4- Full thickness ulceration of the cartilage

SECONDARY OUTCOMES:
cartilage damage measurements | participants will be followed for the duration of the arthrography CT , an expected average of 2 hours
  Quantitative assessment of each location of cartilage damage by maximal diameter in two orthogonal planes tangential to the surface
Image quality (for CBCT and MDCT) | participants will be followed for the duration of the arthrography CT , an expected average of 2 hours
  0 - Insufficient, 1 - Poor, 2 - Average, 3 - Good, 4 - Excellent
Tolerability of the exam (for CBCT and MDCT) | participants will be followed for the duration of the arthrography CT , an expected average of 2 hours
  Perfect, tolerable, hardly tolerable, intolerable
Duration of the exam (for CBCT and MDCT) | participants will be followed for the duration of the arthrography CT , an expected average of 2 hours
  Perfect, tolerable, hardly tolerable, intolerable
Subchondral bone lesion (for CBCT and MDCT) | participants will be followed for the duration of the arthrography CT , an expected average of 2 hours
  No subchondral bone lesion, subchondral bone thickening, subchondral cyst <3mm diameter, subchondral cyst 3 to 5 mm diameter, subchondral cyst >5mm diameter
Lesion of intrinsic ligament (for CBCT and MDCT) | participants will be followed for the duration of the arthrography CT , an expected average of 2 hours
  Yes / No
Osteochondroma (for CBCT and MDCT) | participants will be followed for the duration of the arthrography CT , an expected average of 2 hours
  Each osteochondroma is located (anterior/posterior Medial/ lateral recess, and diameter is measured.: >3mm, 3 to 5 mm, >5mm
Meniscal lesion (for arthrography CBCT and MDCT of the knee) | participants will be followed for the duration of the arthrography CT , an expected average of 2 hours
  No lesion, longitudinal tear, radial tear, complex tear, displaced tear, bucket handle tear

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste PIALAT, MD, Principal Investigator — Hospices Civils de Lyon- Hôpital Edouard Herriot
Locations (1):
- Hospices Civils de Lyon- hôpital Edouard Herriot- service de radiologie pavillon B, Lyon, France

REFERENCES:
- [Result] Debeaupte M, Hermann R, Pialat JB, Martinon A, Truy E, Ltaief Boudrigua A. Cone beam versus multi-detector computed tomography for detecting hearing loss. Eur Arch Otorhinolaryngol. 2019 Feb;276(2):315-321. doi: 10.1007/s00405-018-5214-y. Epub 2018 Nov 23. PMID 30467778